CLINICAL TRIAL: NCT06821217
Title: A Mobile Application as Supportive Treatment of Endometriosis: the Effect on Quality of Life and Endometriosis-associated Pain. A Randomized Controlled Trial.
Brief Title: The Effect of an App-based Intervention on Quality of Life in Patients With Endometriosis.
Acronym: MASQUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-D0105
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis; Pain; Quality of Life; Life Style
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group with histologically confirmed endometriosis (Experimental)
  Interventions: Device: NALU Endo Flow App
- Control group with histologically confirmed endometriosis (No Intervention)
- Intervention group with clinically suspected endometriosis (Experimental)
  Interventions: Device: NALU Endo Flow App
- Control group with clinically suspected endometriosis (No Intervention)

INTERVENTIONS:
Device: NALU Endo Flow App — NALU Endo Flow App is a mobile application for women with endometriosis. The App provides educational information through videos, audios, and texts. Women learn about endometriosis in general with its symptoms, diagnosis, and therapy options such as lifestyle and mindset modification, endometriosis-specific diets, physical and mindfulness exercises. The App includes a diary to track the menstrual cycle and symptoms. Furthermore, access to a WhatsApp community of people with endometriosis is provided and a peer-group call is performed once monthly, as well as one additional monthly Q&A (Question&Answer) call moderated by certified health coaches.
  Arms: Intervention group with clinically suspected endometriosis; Intervention group with histologically confirmed endometriosis

SUMMARY:
The goal of this clinical trial is to learn if an App-based intervention affects the quality of life in patients with suspected or confirmed endometriosis. The main questions it aims to answer are:

* Does the App-based intervention improve the quality of life?
* Does it lead to pain relief? Researchers will compare participants using the App to a control group to see if the App works to improve quality of life and endometriosis-related symptoms.

Participants will:

* Use an App-based intervention or be in the control group (no App-use) for 6 months
* Visit or have a telephone consultation after 3 and 6 months
* Complete a questionnaire to assess the quality of life at inclusion, after 1, 3 and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age 18 or older
* Premenopausal status (menopause is defined as amenorrhea lasting one year or longer)
* Endometriosis, confirmed by surgery or clinically suspected
* Possession of a smartphone

Exclusion Criteria:

* Planned endometriosis surgery or planned hormonal therapy in the study period
* Surgery and/or new hormonal therapy in the last three months
* Malignant diseases
* Pregnancy
* Breastfeeding
* Active desire for pregnancy in the study period
* Fertility treatment
* Simultaneous participation in other intervention studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 308 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Life quality | 6 months
  The primary endpoint will be the change in quality of life in App users assessed by the EHP-30 questionnaire (Endometriosis-Health-Profile-Questionnaire: The questions can be divided into five subscales covering 'pain', 'control and powerlessness', 'social support', 'emotional wellbeing' and 'self-image'. The questionnaire is standardized on a scale from 0 to 100, with lower scores indicating better quality of life.

SECONDARY OUTCOMES:
Pain relief | 6 months
  The secondary endpoint of this study is the change in pain intensity in App users measured by the VAS (Visual Analogue Scale). The VAS is one of various instruments to measure pain intensity. A score of 0 means "no pain", a score of 10 "the worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Gulz, MD, Principal Investigator — University Hospital Bern, Insel Gruppe AG
Locations (1):
- Department of Gynecology and Obstetrics, Women's University Hospital, Inselspital Bern, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No